CLINICAL TRIAL: NCT05311384
Title: Application of a Reimbursable Form of Constraint-Induced Movement Therapy for Upper Extremity Recovery Following Stroke: A Pilot Study
Brief Title: Application of a Reimbursable Form of Constraint-Induced Movement Therapy for Upper Extremity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Sarah dos Anjos, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300008977
Record Dates: First submitted 2022-03-04; First posted 2022-04-05 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: CVA (Cerebrovascular Accident); Stroke; Upper Extremity Paresis
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Keys intervention (Experimental): All participants will receive the Keys CI Therapy protocol over an 8-week intervention period.
  Interventions: Behavioral: Keys Constraint-induced Movement Therapy protocol

INTERVENTIONS:
Behavioral: Keys Constraint-induced Movement Therapy protocol — All participants will receive the Keys CI Therapy protocol over an 8-week intervention period. Specific CI therapy strategies will be delivered, including: 1) supervised movement training will be carried out for 1 hour for 4 days/week for the first 4 weeks, 2 days/week for weeks 5 and 6, and 1 day/week for weeks 7 and 8; 2) participants will use the restraint mitt on their less-affected UE for most of their waking hours for an 8 week period; 3) transfer package methods will be modified to accommodate the longer time period between clinic visits; and 4) participants will be asked to independently perform additional movement training for 30 minutes each day at home.

SUMMARY:
CI therapy is a family of techniques that has systematically applied intensive treatment daily over consecutive days, supervised motor training using a technique called shaping, behavioral strategies to improve the use of the more- affected limb in real life situations called a Transfer Package (TP), and strategies to remind participants to use the more-affected extremity; including restraint of the less-affected arm in the upper extremity (UE) protocol. Numerous studies examining use of CI therapy with UE rehabilitation have demonstrated robust evidence for increasing the amount and the quality of the paretic UE functional use in daily situations of individuals recovering from stroke.

Previous studies have explored the barriers for clinical implementation of the approach, including the amount of time needed by therapists, other resources required and lack of payment for the services. With regards to therapists' time/resources, in the signature CI therapy protocol, therapists supervised movement training for 3 hours daily (except for weekends) for a 12 consecutive-day period. This level of supervision in highly unusual for traditional rehabilitation clinical settings. The treatment schedule is also incompatible with most insurance reimbursement policies in the US. As such, most CI therapy clinics require patients to pay privately with little or no insurance reimbursement. Such practices severely limit the number of patients who can afford to receive CI therapy. Two lines of evidence have suggested that an alternative CI therapy protocol may allow for the essential (or "Key") CI therapy elements to be delivered in a schedule that better utilizes therapist time/resources and is compatible with payment policies of many US insurance companies. One line of evidence comes from findings that indicate that the original 6-hour supervised training schedule could be shortened to as little as 2-hours/daily without a reduction in outcomes. Additional evidence comes from a study exploring the systematic addition and deletion of the signature CI therapy protocol elements indicated that when the transfer package was omitted, outcomes related to functional use were reduced by 50%. These findings were also verified by brain imaging studies conducted concurrently that revealed a much-reduced level of brain remodeling in those not receiving the transfer package. These findings highlight the potential effectiveness of the transfer package and continued movement training by the patient while away from clinical supervision. The hypothesis of this study is that the amount of supervised training could be reduced further and delivered in a distributed schedule (1 to 4 times/ week over an 8-week period) instead of consecutively over a 12-day treatment period. This modification could be possible by adapting and strengthening the transfer package component of the protocol. In order to investigate if all of the Keys intervention protocol is necessary for producing optimal outcomes, the delivery of specific protocol elements will be also explored. Additionally, another round of testing at the 4-week point of the 8-week intervention will be administered to investigate the need for the final 4 weeks of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months after stroke
* Ability to demonstrate minimum movement criteria of more-affected UE including 10 degrees of wrist extension (starting from a fully flexed position), 10 degrees of thumb abduction, and 10 degrees of extension of two additional fingers at all joints
* Score <2.5 on the MAL indicating significant functional deficits of the more-affected UE

Exclusion Criteria:

* Inability to answer the MAL questions and/or provide informed consent
* Score <24 on the Mini-Mental State Examination
* No availability to come to the clinic for the sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Virani SS, Alonso A, Benjamin EJ, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Shay CM, Spartano NL, Stokes A, Tirschwell DL, VanWagner LB, Tsao CW; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2020 Update: A Report From the American Heart Association. Circulation. 2020 Mar 3;141(9):e139-e596. doi: 10.1161/CIR.0000000000000757. Epub 2020 Jan 29. PMID 31992061
- [Background] Taub E, Miller NE, Novack TA, Cook EW 3rd, Fleming WC, Nepomuceno CS, Connell JS, Crago JE. Technique to improve chronic motor deficit after stroke. Arch Phys Med Rehabil. 1993 Apr;74(4):347-54. PMID 8466415
- [Background] Morris DM, Taub E, Mark VW. Constraint-induced movement therapy: characterizing the intervention protocol. Eura Medicophys. 2006 Sep;42(3):257-68. PMID 17039224
- [Background] Pedlow K, Lennon S, Wilson C. Application of constraint-induced movement therapy in clinical practice: an online survey. Arch Phys Med Rehabil. 2014 Feb;95(2):276-82. doi: 10.1016/j.apmr.2013.08.240. Epub 2013 Sep 8. PMID 24025659
- [Background] Viana R, Teasell R. Barriers to the implementation of constraint-induced movement therapy into practice. Top Stroke Rehabil. 2012 Mar-Apr;19(2):104-14. doi: 10.1310/tsr1902-104. PMID 22436358
- [Background] Fleet A, Che M, Mackay-Lyons M, Mackenzie D, Page S, Eskes G, McDonald A, Boyce J, Boe S. Examining the use of constraint-induced movement therapy in canadian neurological occupational and physical therapy. Physiother Can. 2014 Winter;66(1):60-71. doi: 10.3138/ptc.2012-61. PMID 24719511
- [Background] Uswatte G, Taub E, Morris D, Light K, Thompson PA. The Motor Activity Log-28: assessing daily use of the hemiparetic arm after stroke. Neurology. 2006 Oct 10;67(7):1189-94. doi: 10.1212/01.wnl.0000238164.90657.c2. PMID 17030751
- [Background] Morris DM, Uswatte G, Crago JE, Cook EW 3rd, Taub E. The reliability of the wolf motor function test for assessing upper extremity function after stroke. Arch Phys Med Rehabil. 2001 Jun;82(6):750-5. doi: 10.1053/apmr.2001.23183. PMID 11387578
- [Background] Duncan PW, Wallace D, Lai SM, Johnson D, Embretson S, Laster LJ. The stroke impact scale version 2.0. Evaluation of reliability, validity, and sensitivity to change. Stroke. 1999 Oct;30(10):2131-40. doi: 10.1161/01.str.30.10.2131. PMID 10512918
- [Background] ZUNG WW. A SELF-RATING DEPRESSION SCALE. Arch Gen Psychiatry. 1965 Jan;12:63-70. doi: 10.1001/archpsyc.1965.01720310065008. No abstract available. PMID 14221692
- [Background] Toomey M, Nicholson D, Carswell A. The clinical utility of the Canadian Occupational Performance Measure. Can J Occup Ther. 1995 Dec;62(5):242-9. doi: 10.1177/000841749506200503. PMID 10152880
- [Background] Wolf SL, Winstein CJ, Miller JP, Thompson PA, Taub E, Uswatte G, Morris D, Blanton S, Nichols-Larsen D, Clark PC. Retention of upper limb function in stroke survivors who have received constraint-induced movement therapy: the EXCITE randomised trial. Lancet Neurol. 2008 Jan;7(1):33-40. doi: 10.1016/S1474-4422(07)70294-6. PMID 18077218
- [Background] Morris DM, Taub E, Macrina DM, Cook EW, Geiger BF. A method for standardizing procedures in rehabilitation: use in the extremity constraint induced therapy evaluation multisite randomized controlled trial. Arch Phys Med Rehabil. 2009 Apr;90(4):663-8. doi: 10.1016/j.apmr.2008.09.576. PMID 19345784
- [Background] Andrabi M, Taub E, Mckay Bishop S, Morris D, Uswatte G. Acceptability of constraint induced movement therapy: influence of perceived difficulty and expected treatment outcome. Top Stroke Rehabil. 2022 Oct;29(7):507-515. doi: 10.1080/10749357.2021.1956046. Epub 2021 Aug 23. PMID 34425065
- [Background] Taub E, Uswatte G, Mark VW, Morris DM. The learned nonuse phenomenon: implications for rehabilitation. Eura Medicophys. 2006 Sep;42(3):241-56. PMID 17039223
- [Background] Uswatte G, Taub E, Morris D, Barman J, Crago J. Contribution of the shaping and restraint components of Constraint-Induced Movement therapy to treatment outcome. NeuroRehabilitation. 2006;21(2):147-56. PMID 16917161
- [Background] Shi YX, Tian JH, Yang KH, Zhao Y. Modified constraint-induced movement therapy versus traditional rehabilitation in patients with upper-extremity dysfunction after stroke: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2011 Jun;92(6):972-82. doi: 10.1016/j.apmr.2010.12.036. PMID 21621674
- [Background] Taub E, Uswatte G, Mark VW, Morris DM, Barman J, Bowman MH, Bryson C, Delgado A, Bishop-McKay S. Method for enhancing real-world use of a more affected arm in chronic stroke: transfer package of constraint-induced movement therapy. Stroke. 2013 May;44(5):1383-8. doi: 10.1161/STROKEAHA.111.000559. Epub 2013 Mar 21. PMID 23520237
- [Derived] Dos Anjos S, Bowman M, Morris D. Effects of a Distributed Form of Constraint-Induced Movement Therapy for Clinical Application: The Keys Treatment Protocol. Brain Sci. 2025 Jan 17;15(1):87. doi: 10.3390/brainsci15010087. PMID 39851454

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Despite the various strategies were used for recruitment such as reaching out to outpatient clinics in our area, posting recruitment flyer in social media pages, attending stroke support groups, including clinicians and rehabilitation professionals of the stroke unit of our institution, and contacting participants from other studies conducted by the authors, the final sample was smaller than anticipated. The initial sample of 14 was reduced to 10 to follow the funding source timeline.
Pre-assignment Details: All participants received the same intervention, thus all individuals were assigned to the same group.
Period: Overall Study
Arm/Group | Keys Intervention
Started | 10
Completed | 7
Not Completed | 3
Not completed — Uncontrolled health conditions | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Keys Intervention
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 61.7 [46 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/Black | 4
  White | 6
Region of Enrollment [Number; unit: participants]
  United States | 10
Type of stroke [Count of Participants; unit: Participants]
  Ischemic | 5
  Hemorrhagic | 2
  Unsure | 3
Time since onset [Mean (Full Range); unit: months] | 26.9 [6 to 56]
Affected side [Count of Participants; unit: Participants]
  Left | 5
  Right | 5
Pre-Morbid Handedness [Count of Participants; unit: Participants]
  Right | 8
  Left | 2

OUTCOME MEASURES:

1. Primary Outcome: Motor Activity Log (MAL)
Description: The MAL assesses how much and how well the individuals uses the affected upper extremity in 30 different daily activities. It will be used to investigate the change in spontaneous use of the affected upper extremity comparing the scores collected before and in the middle of the treatment. The MAL includes two scales: Amount of use (AOU) and Quality of Movement (QOM) and each one of them is scored from 0-10, and higher scores denote more frequent spontaneous use and better quality of movement of the affected arm.
Time Frame: Pre-treatment
Measure: Mean (Full Range); unit: Points
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
Points
  Amount of Use (AOU) Scale | 1 [0.3 to 1.6]
  Quality of Movement (QOM) | 1.1 [0.3 to 1.5]

2. Primary Outcome: Motor Activity Log (MAL)
Description: as for outcome 1
Time Frame: 4 weeks after starting the intervention (middle of the protocol)
Measure: Mean (Full Range); unit: Points
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
Points
  Amount of Use (AOU) Scale | 3.5 [1.9 to 4.5]
  Quality of Movement (QOM) | 3.3 [2.0 to 4.4]

3. Primary Outcome: Motor Activity Log (MAL)
Description: The MAL assesses how much and how well the individuals uses the affected upper extremity in 30 different daily activities. It will be used to investigate the change in spontaneous use of the affected upper extremity comparing the scores collected before and in the middle of the treatment.The MAL assesses how much and how well the individuals uses the affected upper extremity in 30 different daily activities. It will be used to investigate the change in spontaneous use of the affected upper extremity before and after the treatment. The assessment is scored from 0-10, and higher scores denote more frequent spontaneous use and quality of movement of the affected arm.
Time Frame: after the intervention (8 weeks after starting the protocol)
Measure: Mean (Full Range); unit: Points
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
Points
  Amount of Use (AOU) | 3.9 [2.5 to 4.8]
  Quality of Movement (QOM) | 3.4 [1.7 to 4.7]

4. Primary Outcome: Motor Activity Log (MAL)
Description: as for outcome 1
Time Frame: 3 months after the end of the treatment.
Measure: Mean (Full Range); unit: Points
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
Points
  Amount of Use (AOU) | 4.0 [2.8 to 4.8]
  Quality of Movement | 3.7 [2.1 to 4.8]

5. Primary Outcome: Canadian Occupational Performance Measure (COPM)
Description: The COPM is a self-reported measure regarding the individual's occupational performance in self-care, productivity, and leisure activities. The COPM will be administered to explore the changes in occupational performance comparing the scores collected before, in the middle of the treatment and after the treatment. Five of the activities considered more important to the individuals are scored through two different scales: the performance and the satisfaction scales. Each one is scored from 0-10, and higher scores denote higher satisfaction, and quality of performance.
Time Frame: Pre-treatment
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
Score on a scale
  Performance | 1.9 [1 to 3]
  Satisfaction | 1.3 [1 to 1.4]

6. Primary Outcome: Canadian Occupational Performance Measure (COPM)
Description: as for outcome 5
Time Frame: 4 weeks after starting the intervention (middle of the protocol)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale
  Performance | 5.5 [3.8 to 7.6]
  Satisfaction | 4.7 [1.6 to 6]

7. Primary Outcome: Canadian Occupational Performance Measure (COPM)
Description: as for outcome 5
Time Frame: after the intervention (8 weeks after starting the protocol)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale
  Performance | 6.3 [3.8 to 8.4]
  Satisfaction | 6.1 [3.2 to 8.8]

8. Primary Outcome: Canadian Occupational Performance Measure (COPM)
Description: as for outcome 5
Time Frame: 3 months after the end of the treatment.
Population: The administration of the COPM was included in the 3 month follow up assessment visit after the study has started. With the delay in having this modification approved by the institutional ethics committee, the the first two participants did not have COPM administered in the follow up visit. Therefore, data from 5 out of the 7 participants in this study are reported here.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 5
score on a scale
  Performance | 6.6 [3 to 9.2]
  Satisfaction | 6.1 [1.4 to 9.4]

9. Primary Outcome: Wolf Motor Function Test (WMFT) - Performance Time
Description: The WMFT measures upper extremity motor function in terms of quality of movement and performance time. The WMFT will be administered to investigate changes in motor function of the affected arm comparing the scores collected before and in the middle of the treatment. The WMFT is scored in two different ways: through performance times (in seconds) and quality of performance through the Functional Ability Scale (FAS). The FAS ranges from 0-5, in which 0 represents inability to perform the task, and 5 is given for performances close o before the stroke. The tasks are also timed with a stopwatch and lower performance time denotes better motor function.
Time Frame: Pre-treatment
Measure: Median (Full Range); unit: seconds
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
seconds | 5.32 [3.17 to 10.64]

10. Primary Outcome: Wolf Motor Function Test (WMFT) - Performance Time
Description: as for outcome 9
Time Frame: 4 weeks after starting the intervention (middle of the protocol)
Measure: Median (Full Range); unit: Seconds
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
Seconds | 5.32 [3.17 to 10.64]

11. Primary Outcome: Wolf Motor Function Test (WMFT) - Performance Time
Description: as for outcome 9
Time Frame: after the intervention (8 weeks after starting the protocol)
Measure: Median (Full Range); unit: Seconds
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
Seconds | 3.82 [2.43 to 31.26]

12. Primary Outcome: Wolf Motor Function Test (WMFT) - Functional Ability Scale
Description: as for outcome 9
Time Frame: Pre-treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale | 3 [2 to 3.5]

13. Primary Outcome: Wolf Motor Function Test (WMFT) - Functional Ability Scale
Description: as for outcome 9
Time Frame: 4 weeks after starting the intervention (middle of the protocol)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale | 3 [2 to 3.5]

14. Primary Outcome: Wolf Motor Function Test (WMFT) - Functional Ability Scale
Description: as for outcome 9
Time Frame: after the intervention (8 weeks after starting the protocol)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale | 3 [2 to 4]

15. Secondary Outcome: Stroke Impact Scale (SIS)
Description: The SIS is a self-reported measure of disability and quality of life after stroke. The SIS will be administered to investigate changes in quality of life comparing the scores collected before and in the middle of the treatment. The SIS includes 9 domains and each one of them ranges from 0-100, where lower score mean more difficulty performing the task and lower self-perceived recovery. The domains are: 1) Strength, 2) Memory; 3) Mood; 4) Communication; 5) Activities of Daily Living (ADLs)/ Instrumental ADLs (IADLs); 6) Mobility; 7) Hand Function; 8) Participation; and 9) Recovery.
Time Frame: Pre-treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale
  Strength | 51.8 [25 to 75]
  Memory | 59.8 [38.1 to 85.7]
  Mood | 64.2 [50 to 69.4]
  Communication | 90.5 [46.4 to 100]
  ADLs / IADLs | 56.8 [55 to 90]
  Mobility | 77 [47.2 to 100]
  Hand Function | 36.1 [25 to 75]
  Participation | 56.4 [25 to 81.3]
  Recovery | 58.9 [35 to 80]

16. Secondary Outcome: Stroke Impact Scale (SIS)
Description: as for outcome 15
Time Frame: 4 weeks after starting the intervention (middle of the protocol)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale
  Strength | 59.8 [31.3 to 87.5]
  Memory | 63.9 [35.7 to 66.7]
  Mood | 63.9 [55.6 to 69.4]
  Communication | 91.8 [60.7 to 100]
  ADLs / IADLs | 70.4 [40 to 92.5]
  Mobility | 79.4 [33.4 to 97.2]
  Hand function | 60.7 [10 to 90]
  Participation | 69.6 [25 to 93.8]
  Recovery | 59.3 [30 to 85]

17. Secondary Outcome: Stroke Impact Scale (SIS)
Description: as for outcome 15
Time Frame: after the intervention (8 weeks after starting the protocol)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale
  Strength | 65.2 [43.8 to 87.5]
  Memory | 61.6 [38.1 to 100]
  Mood | 65.5 [58.3 to 69.4]
  Communication | 90.3 [50 to 100]
  ADLs / IADLs | 77.1 [50 to 97.5]
  Mobility | 82.9 [44.4 to 100]
  Hand Function | 65 [30 to 90]
  Participation | 75 [43.8 to 100]
  Recovery | 70 [35 to 85]

18. Secondary Outcome: Stroke Impact Scale (SIS)
Description: as for outcome 15
Time Frame: 3 months after the end of the treatment.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale
  Strength | 65.2 [25 to 81.3]
  Memory | 67.7 [52.4 to 100]
  Mood | 69 [63.9 to 75]
  Communication | 93.4 [60.7 to 100]
  ADLs / IADLs | 81.1 [60 to 97.5]
  Mobility | 84.1 [66.7 to 100]
  Hand Function | 70.7 [30 to 100]
  Participation | 76.8 [37.5 to 100]
  Recovery | 76.4 [60 to 90]

19. Secondary Outcome: Zung Self-Rating Depression Scale
Description: The ZDS is a self-reported outcome that measures the presence of specific symptoms related to depression. The final score ranges from 20-80, where scores are classified as normal (<50), mild depression (50 to 59), moderate to marked major depression (60 to 69), and severe to extreme major depression (>70). The ZDS will be administered to investigate changes in depressive symptoms comparing the scores collected before and in the middle of the treatment.
Time Frame: Pre-treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale | 34.1 [26 to 45]

20. Secondary Outcome: Zung Self-Rating Depression Scale
Description: as for outcome 19
Time Frame: 4 weeks after starting the intervention (middle of the protocol)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale | 32.1 [25 to 49]

21. Secondary Outcome: Zung Self-Rating Depression Scale
Description: The ZDS is a self-reported outcome that measures the presence of specific symptoms related to depression. The ZDS is a self-reported outcome that measures the presence of specific symptoms related to depression. The final score ranges from 20-80, where scores are classified as normal (<50), mild depression (50 to 59), moderate to marked major depression (60 to 69), and severe to extreme major depression (>70). The ZDS will be administered to investigate changes in depressive symptoms comparing the scores collected before and after the treatment.
Time Frame: after the intervention (8 weeks after starting the protocol)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale | 30.4 [24 to 49]

22. Secondary Outcome: Zung Self-Rating Depression Scale
Description: The ZDS is a self-reported outcome that measures the presence of specific symptoms related to depression. The ZDS is a self-reported outcome that measures the presence of specific symptoms related to depression. The final score ranges from 20-80, where scores are classified as normal (<50), mild depression (50 to 59), moderate to marked major depression (60 to 69), and severe to extreme major depression (>70). The ZDS will be administered to investigate changes in depressive symptoms comparing the scores collected right after of the treatment and 3 months after the end of the treatment.
Time Frame: 3 months after the end of the treatment.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Keys Intervention
Number analyzed (Participants) | 7
score on a scale | 31 [22 to 44]

ADVERSE EVENTS:
Time Frame: Adverse events information were monitored and collected throughout the eight weeks of intervention. All participants were asked about soreness and fatigue at the beginning of each treatment session.
Description: The definition of the adverse events from clinicaltrials.gov was followed in this study.
Arm/Group | Keys Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
This study has a small sample size due to challenges in recruitment and enrollment. The recruitment process was somewhat impacted by the COVID-19 pandemic due to transportation limitations, and difficulties in controlling health conditions (e.g., arterial hypertension). While the results of this pilot trial are promising, larger studies with comparison groups are needed. Additionally, the use of wearable sensors that could provided data comparable to the MAL scores would be indicated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT05311384/Prot_SAP_ICF_000.pdf